CLINICAL TRIAL: NCT05285618
Title: Predicting the Perceptual Experience of Argus II Retinal Prosthesis System Users
Brief Title: The Perceptual Experience of Argus II Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Santa Barbara (Other)
Collaborators: Johns Hopkins University (Other); University of Michigan (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Michael Beyeler, PhD, Professor, University of California, Santa Barbara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R00EY029329 (NIH); R00EY029329 (NIH)
Record Dates: First submitted 2022-02-04; First posted 2022-03-17 (Actual); Results first posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Argus II users (Experimental): This Basic Experimental Studies Involving Humans (BESH) study investigates phosphene perception and performance factors in blind participants implanted with the Argus II retinal prosthesis system. Using paired-electrode stimulation, we analyze how phosphene shape and number are influenced by neuroanatomical factors, stimulus parameters, and spatial offsets. Additionally, we examine the causes of high current thresholds and limited spatial resolution, which impede pattern vision in Argus II devices. This research aims to provide insights for optimizing stimulation strategies and improving retinal prosthesis design.
  Interventions: Device: Argus II

INTERVENTIONS:
Device: Argus II — Participants used the Argus II retinal prosthesis system in both experiments to perform visual perception tasks.

SUMMARY:
This Basic Experimental Studies Involving Humans (BESH) study investigates phosphene perception and performance factors in blind participants implanted with the Argus II retinal prosthesis system. Using paired-electrode stimulation, we analyze how phosphene shape and number are influenced by neuroanatomical factors, stimulus parameters, and spatial offsets. Additionally, we examine the causes of high current thresholds and limited spatial resolution, which impede pattern vision in Argus II devices. This research aims to provide insights for optimizing stimulation strategies and improving retinal prosthesis design.

DETAILED DESCRIPTION:
This study focuses on two experiments involving blind participants implanted with the Argus II retinal prosthesis:

Experiment 1: Paired-Electrode Phosphene Perception The study retrospectively analyzes 3548 phosphene drawings made by three participants. We investigate the impact of single- and paired-electrode stimulation on phosphene shape (area, perimeter, major/minor axis length) and the number of perceived phosphenes. Neuroanatomical parameters, including electrode-retina distance, electrode-fovea distance, and electrode-electrode distance (both along-axon and between-axon), are correlated with these outcomes. Statistical analyses include linear regression and partial correlation to examine the relationship between stimulation parameters and phosphene perception.

Experiment 2: Performance Factors in Argus II Prostheses This study explores the factors contributing to high current amplitude thresholds and poor spatial resolution in three participants. We measure current amplitude thresholds and two-point discrimination (the ability to distinguish stimulation on one versus two electrodes). Data from psychophysical experiments and simulations are analyzed to identify the roles of axonal stimulation, electrode lift, and retinal damage in limiting device performance.

These experiments aim to advance the understanding of epiretinal stimulation and inform the development of future retinal prostheses with improved spatial resolution and sensitivity.

ELIGIBILITY:
Inclusion criteria:

* Subject must be at least 25 years of age;
* Subject has been implanted with the Argus II system;
* Subject's eye has healed from surgery and the surgeon has cleared the subject for programming;
* Subject has the cognitive and communication ability to participate in the study (i.e., follow spoken directions, perform tests, and give feedback);
* Subject is willing to conduct psychophysics testing up to 4-6 hours per day of testing on 3-5 consecutive days;
* Subject is capable of understanding patient information materials and giving written informed consent;
* Subject is able to walk unassisted.

Exclusion criteria:

* Subject is unwilling or unable to travel to testing facility for at least 3 days of testing within a one-week timeframe;
* Sighted controls: Subject has a history of motion sickness or flicker vertigo
* Subject does not speak English;
* Subject has language or hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Beyeler, PhD, Principal Investigator — University of California, Santa Barbara
Locations (3):
- United States (3):
  - University of California, Santa Barbara, Santa Barbara, California
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available from the investigative team, following initial publication of the results
Supporting Information: Study Protocol, SAP
Time Frame: Spring 2023 onward
Access Criteria: Any researchers with a legitimate reason for wishing to re-analyze the data or compare them to study data collected in similar experiments

REFERENCES:
- [Result] Yucel EI, Sadeghi R, Kartha A, Montezuma SR, Dagnelie G, Rokem A, Boynton GM, Fine I, Beyeler M. Factors affecting two-point discrimination in Argus II patients. Front Neurosci. 2022 Aug 24;16:901337. doi: 10.3389/fnins.2022.901337. eCollection 2022. PMID 36090266
- [Result] Hou Y, Nanduri D, Granley J, Weiland JD, Beyeler M. Axonal stimulation affects the linear summation of single-point perception in three Argus II users. J Neural Eng. 2024 Apr 8;21(2):026031. doi: 10.1088/1741-2552/ad31c4. PMID 38457841

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Argus II Users
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Argus II Users: Blind individuals previously implanted with the Argus II retinal prosthesis system participated in two experiments. The first experiment tested phosphene perception by varying the spatial offsets and temporal delays between pairs of electrodes. The second experiment tested the effect of gamification on circle localization and motion discrimination tasks.
  Argus II: Participants used the Argus II retinal prosthesis system in both experiments to perform visual perception tasks.
  Gamification: Participants performed gamified versions of circle localization and motion discrimination tasks designed to improve engagement and task performance.
Arm/Group | Argus II Users
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Phosphenes Perceived
Description: Number of phosphenes perceived in response to paired-electrode stimulation across 5 spatial distances and 7 temporal interpulse delays. Phosphenes are brief sensations of light or visual flashes that occur in the absence of an external light source. A response is counted as a phosphene if the participant reports any visual sensation consistent with a flash of light.
Time Frame: during single-session testing
Population: Data were collected in 6 participants ranging in age from 45 to 88 years old. One participant was female. All identified as white, non-hispanic.
Measure: Mean (Standard Deviation); unit: number of phosphenes
Groups:
- Argus II Users: Blind individuals previously implanted with the Argus II retinal prosthesis system were invited to join the study.
Arm/Group | Argus II Users
Number analyzed (Participants) | 6
number of phosphenes
  Delay 0 | 1.09 (0.910)
  Delay 4ms | 1.43 (0.555)
  Delay 12ms | 1.46 (0.538)
  Delay 29ms | 1.41 (0.570)
  Delay 50ms | 1.48 (0.511)
  Delay 178ms | 1.37 (0.544)
  Delay 419ms | 1.36 (0.639)
  Distance (808 - 1834um) | 1.24 (0.642)
  Distance (1835 - 2856um) | 1.44 (0.685)
  Distance (2857 - 3877um) | 1.31 (0.622)
  Distance (3878 - 4898um) | 1.41 (0.663)
  Distance (4899 - 5920um) | 1.45 (0.631)
Statistical Analysis 1: Comparison: Argus II Users; The model tested whether stimulation delay ('abs_delay'), retinal distance ('dist_ret'), and their interaction ('abs_delay:dist_ret') affect the number of elicited phosphenes ('num_phosphenes'); Test type: Other — A linear mixed model accounted for repeated measures ('subject_id' as a random factor). No power calculation was performed, but the sample size (1,485 observations, 6 subjects) supports robust estimation; p = 0.002, Mixed Models Analysis — P-values are unadjusted for multiple comparisons, as the analysis focused on a limited number of predictors. The a priori threshold for statistical significance was set at p<0.05; We hypothesize that the parameter 'dist_ret' may influence the number of phosphenes perceived ('num_phosphenes'), while the roles of 'abs_delay' and its interaction with 'dist_ret' may be less pronounced. Further evaluation of these parameters will be conducted in the Results section

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Argus II Users
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT05285618/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT05285618/SAP_001.pdf
  • Informed Consent Form (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT05285618/ICF_002.pdf